CLINICAL TRIAL: NCT06763679
Title: Comparative Effects of Spencer Technique With and Without Acromioclavicular Mobilization on Pain, Range of Motion and Functional Disability Among Patients of Frozen Shoulder
Brief Title: Compare the Effect of Spencer Technique With and Without AC Mobilization for FS Pathients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0126
Record Dates: First submitted 2025-01-01; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Frozen
Keywords: Spencer Technique; Acromioclavicular joint; Mobilization; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobilization (Experimental): Spencer Technique with Acromioclavicular mobilization
  Interventions: Other: mobilization
- Traditional physical therapy (Active Comparator): Spencer technique
  Interventions: Other: traditional physical therapy

INTERVENTIONS:
Other: mobilization — Acromioclavicular joint mobilization:
  * The patient is placed in the supine position and the upper limb is placed in a physiological position with the patient's arm clinging to the body and the hand on the abdomen, which causes the capsule to stretch less and the technique to be less painful.
  * The therapist placed the tips of his both thumbs on the anterior surface of the clavicle adjacent to the ACJ and spread his other fingers out for stability and his forearm was situated in line with the posterior movement at the ACJ.
  * ACJ mobilization was performed in up to 30-minute individual sessions by a single trained therapist.
  * The treatment techniques were anterior to posterior passive accessory glides of the distal end of the clavicle categorized from Grade III
  * Grade III is used at a large amplitude from the middle of the joint ROM to the start of the constraint. Grade III will apply for stimulating a stretching to relieve joint stiffness in a shorter tissue
  Arms: mobilization
Other: traditional physical therapy — Spencer technique:
  * The patient was resting on their side, with the affected shoulder raised.
  * In 7 separate movements, the therapist used the proximal hand to stabilize the shoulder girdle, while the distal hand applied force to the restrictive barrier of the shoulder.
  * Shoulder extension, circumduction with compression, shoulder flexion, circumduction with distraction, abduction, adduction with internal rotation, and glenohumeral pump were the exercises performed.
  * The patients were advised to employ their muscle energy technique against the small resistance provided by the therapist for 3-5 seconds throughout each movement.
  * Over the course 5 days a week, the exercise was repeated 3-5 times per session, with rest breaks.
  Arms: Traditional physical therapy

SUMMARY:
The propose of the study will help the clinicians provide an evidence-based approach for the application of Spencer technique and acromioclavicular mobilization, an application of these techniques on pain, range of motion and functional disability of patients of frozen shoulder. So, that it can be determined which treatment is superior in terms of achieving better results in the management regime.

DETAILED DESCRIPTION:
A case report to determine an Integrated Physical Therapy Using Spencer Technique in the Rehabilitation of a Patient With a Frozen Shoulder (FS). In this case report, the 57 years old male occupation of shopkeeper came with the complaint of right frozen shoulder. The treatment of Spencer's Technique with stathe study in 2023 about Acromioclavicular joint mobilizations for the management of grade I sternoclavicular joint sprain. In this case report, after sustaining a grade I posteriorly directed sternoclavicular sprain in a car accident, the patient, a 34-year-old woman, had five sessions of acromioclavicular joint mobilizations and rehabilitative exercise for her shoulder complex over a period of six weeks. The result was that a combination of acromioclavicular joint mobilizations and therapeutic exercise was suitable conservative management for grade I sternoclavicular sprainndard management was given for 3 weeks. The SPADI questionnaire was used. It was concluded that the Spencer Technique had a significant effect on reducing pain, increase shoulder range of motion and improve functional disability.

in 2023 about Prevelence of musculoskeletal disorders in medical laboratory technicians. The 22 years old patient came with complaint of pain in right shoulder during overhead sports activities. The test for impingement like empty can test, Neer's impingement test, Hawkins Kenneddy test was positive. The patient treated with Spencer technique. It was concluded that the Spencer Technique was effective for shoulder impingement syndrome to increase range of motion.

An experimental study in 2023 about comparative effect of gong's mobilization and Spencer technique to manage frozen shoulder. In this study, there were 30 subjects which diagnosed with unilateral frozen shoulder were randomized into 2 groups by simple random method. The group 1 received Spencer technique with ultrasound and Codman's pendulum exercise and group 2 received gong's mobilization with ultrasound and Codman's pendulum exercise. The conclusion was that gong's mobilization was more effective than Spencer technique with ultrasound and Codman's pendulum exercises in treating frozen shoulder patients.

A quasi experimental study about the immediate effect of acromioclavicular joint mobilization on shoulder range of motion. In this study, 30 healthy participants were taken with a complaint of decrease range of motion. The participants received acromioclavicular joint mobilization The result was that acromioclavicular joint mobilization increase the shoulder range of motion.

A randomized controlled trial in 2022 about Spencer muscle energy technique versus conventional treatment in frozen shoulder. In this study, the 60 participants with idiopathic frozen shoulder were examined and only 40 were received the treatment and randomly divided into 2 groups. The first group took the treatment of spencer muscle energy technique and second group received conventional treatment. This study concluded that spencer muscle energy technique was more beneficial for reducing pain in shoulder as well as conventional treatment improve range of motion.

A randomized clinical trial was conducted about Effectiveness of acromioclavicular joint mobilization and physical therapy vs physical therapy alone in patients with frozen shoulder in 2021. In this study, there were two groups: an experimental group and control group. The experimental group got acromioclavicular joint mobilization and physical therapy but control group contain only physical therapy. The result was that acromioclavicular joint mobilization with physical therapy treatment was more effective to increase range of motion, decrease pain and disability.

In 2020, a single blind randomized control trial was conducted about comparison of spencer muscle energy technique and passive stretching in adhesive Capsulitis. There were 60 patients participated in this study. All patients are randomly divided into two groups: group 1 received spencer muscle energy technique and group 2 received passive stretching. The study was concluded that the spencer technique used in group 1 was more effectual than passive stretching used in group 2.

Comparing Spencer technique with and without Acromioclavicular mobilization in patients with frozen shoulder lies in the integration of specific techniques, the focus on a distinct patient population, and the comprehensive assessment of pain, range of motion, and functional disability. The study has the potential to advance our understanding of effective interventions for frozen shoulder and inform evidence-based practices in rehabilitation and physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female both are included
* Age of 50-60 years
* Unilateral frozen shoulder stage 2 with pain lasting for more than 1 month
* Capsular pattern of motion restriction (lateral rotation, abduction, medial rotation)
* More than 50% loss of passive movement of shoulder

Exclusion Criteria:

* Rotator cuff tear
* Dislocation of shoulder
* Shoulder subluxation
* Upper limb fracture
* History of shoulder surgery
* All other co-morbidities are excluded

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-01-13 (Estimated); Study Completion 2025-01-13 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index | 6th week
  SPADI is one of the most often used PROMs to evaluate pain and impairment in individuals with frozen shoulder. When used to measure shoulder problems, SPADI has demonstrated exceptional construct validity and reliability, primarily in patients who come with shoulder discomfort at the primary care level. The SPADI was created to assess the extent of shoulder pain and discomfort during everyday activities by the patients themselves. There are 13 components total, with 5 related to pain and 8 related to disability, components were rated using a visual analog scale. The responses are added up and converted into a composite score of 100, where 100 represents the highest level of shoulder discomfort and disability and zero represents the lowest level.

SECONDARY OUTCOMES:
universal goniometer | 6th week
  The measurement of joint range of motion (ROM) is an essential procedure used in physical therapy, known as goniometry(22).
  Goniometry, the measurement of joint angles, traditionally performed with a universal goniometer (UG), is a commonly utilized assessment tool in monitoring problems of the musculoskeletal system, as well as the progression of rehabilitation interventions.
numeric pain rating scale | 6th week
  Numeric Pain Rating Scale (NRS-11), which is an eleven-point scale in which the end points are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10). NPRS-11 pain severity score of "4" is frequently given special significance in this regard, suggesting it as a potential threshold value for pain severity in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Humera mubashar, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Bajwa hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phansopkar P, Qureshi MI. An Integrated Physical Therapy Using Spencer's Technique in the Rehabilitation of a Patient With a Frozen Shoulder: A Case Report. Cureus. 2023 Jun 30;15(6):e41233. doi: 10.7759/cureus.41233. eCollection 2023 Jun. PMID 37529524